CLINICAL TRIAL: NCT01413529
Title: HEART to HAART: Smartphone Intervention to Improve HAART Adherence for Drug Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Seth Himelhoch, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: HP-00049374; 1R34DA032411 (NIH)
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: HIV; Drug Use Disorders
Keywords: HIV infected persons with co-occurring drug use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HEART to HAART (Experimental): HEART to HAART intervention is designed to enhance ongoing adherence counseling by providing (1) real time information about medication adherence (using Wisepill device); (2) periodic assessment of medication side effects, depressive symptoms and drug use frequency (as these are linked to poor adherence among drug users) using ecological momentary assessment and (3) tailored education, recommendation and encouragement based on assessments. The participant (using their phone) and their adherence team (using a clinician interface) can jointly track real time changes in adherence increasing the potential for shared decision-making.
  Interventions: Behavioral: HEART to HAART
- Adherence counseling (Active Comparator): Adherence counseling with the addition of a smart phone control
  Interventions: Behavioral: adherence counseling with the addition of smartphone control

INTERVENTIONS:
Behavioral: HEART to HAART — The HEART to HAART intervention is designed to enhance ongoing adherence counseling by providing (1) real time information about medication adherence (using Wisepill device); (2) periodic assessment of medication side effects, depressive symptoms and drug use frequency (as these are linked to poor adherence among drug users) using ecological momentary assessment and (3) tailored education, recommendation and encouragement based on assessments. The participant (using their phone) and their adherence team (using a clinician interface) can jointly track real time changes in adherence increasing the potential for shared decision-making.
  Arms: HEART to HAART
Behavioral: adherence counseling with the addition of smartphone control — Participants will receive adherence counseling with the addition of smartphone control.
  Arms: Adherence counseling

SUMMARY:
HIV infected drug users have greater difficulty adhering to highly active antiretroviral therapy compared to non-drug users. As sustained adherence to highly active antiretroviral therapy is critical to reducing HIV related morbidity, mortality, and reducing the spread of HIV, innovative and potentially sustainable treatment strategies that can optimize the durability of adherence enhancing interventions among drug users is urgently needed. The goal of this study is to further develop and pilot test a smartphone based intervention called HEART (Helping Enhance Adherence to Retroviral therapy using Technology) to HAART, to enhance adherence to HAART among HIV infected drug users.

DETAILED DESCRIPTION:
Significance: HIV infected drug users have greater difficulty adhering to HAART compared to non-drug users. As sustained adherence is critical to reducing HIV related morbidity and mortality, innovative and potentially sustainable treatment strategies that can optimize the durability of adherence enhancing interventions among drug users are urgently needed. Increasingly, interventions using communication technologies (e.g.,smartphones) to assess and enhance treatments are being used for a variety of somatic, mental health and substance abuse conditions.

Innovation/Approach: Consistent with the National Institute on Drug Abuse's mission to develop novel technological based interventions to promote adherence to HAART the goal of this study is to use the stage model of behavioral therapy research to adapt, further develop, complete preliminary usability and pilot testing of a smart phone based intervention called HEART (Helping Enhance Adherence to Retroviral therapy using Technology) to HAART, to enhance, promote, and improve long-term adherence to HAART among HIV infected drug users in the non-methadone maintenance setting. Informed by Wagner's Chronic Care Model, the HEART to HAART intervention is designed to enhance ongoing adherence counseling by providing (1) real time information about medication adherence (using Wisepill device); (2) periodic assessment of medication side effects, depressive symptoms and drug use frequency (as these are linked to poor adherence among drug users) using ecological momentary assessment and (3) tailored education, recommendation and encouragement based on assessments. The participant (using their phone) and their adherence team (using a clinician interface) can jointly track real time changes in adherence increasing the potential for shared decision-making.

This proposal has three aims consistent with stage 1A and 1B of the stage of behavioral therapy research. Aims 1 and 2 seek to adapt and further develop (Stage 1A) HEART to HAART. Aims 1 and 2 will use an iterative user-centered design that allows end users of a system to influence how a design takes shape to increase the ease with which a system can be learned and used. Aim 3 will test the preliminary efficacy (Stage 1B) of the finalized form of HEART to HAART. In aim 3, a total of 50 HIV infected, drug users receiving adherence counseling at an urban, outpatient HIV clinic will be randomly assigned to receive either HEART to HAART versus usual care with the addition of a smart phone control. The intervention will last 24 weeks and the primary outcome will be change in adherence as measured by unannounced telephone based random pill counts. Changes in biological outcomes including HIV viral load and CD4 count will also be evaluated.

Implication: If shown to be acceptable and efficacious HEART to HAART may introduce a fundamentally new method of HAART medication self-management and provide a tailored, potentially sustainable and less cost intensive intervention that can increase adherence among HIV infected drug users over the long term.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV
* English speaking
* History of drug use in the last 6 months
* Able to carry a cell phone
* Able to read English
* Starting or switching to a new anti-retroviral medications
* Receiving care in a clinic participating in the study

Exclusion Criteria:

* Clinical problems that would not allow someone to use a cell phone or fulfill study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
adherence to antiretroviral medication | 6 months
  telephone based unannounced pill counts

CONTACTS AND LOCATIONS:
Overall Officials: Seth Himelhoch, MD, MPH, Principal Investigator — University of Maryland
Locations (1):
- Jacques Initiative, Baltimore, Maryland, United States